CLINICAL TRIAL: NCT00753688
Title: A Randomized Double Blind Phase III Trial of Pazopanib Versus Placebo in Patients With Soft Tissue Sarcoma Whose Disease Has Progressed During or Following Prior Therapy
Brief Title: Pazopanib Versus Placebo in Patients With Soft Tissue Sarcoma Whose Disease Has Progressed During or Following Prior Therapy
Acronym: PALETTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VEG110727; NCT00794521 (obsolete NCT alias)
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Sarcoma, Soft Tissue
Keywords: metastatic soft-tissue sarcoma; pazopanib; Soft Tissue Sarcoma; placebo
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLACEBO (Placebo Comparator): matching placebo 800 mg once daily orally
  Interventions: Drug: Placebo
- PAZOPANIB (Experimental): 800 mg once daily orally
  Interventions: Drug: PAZOPANIB

INTERVENTIONS:
Drug: PAZOPANIB — 800 mg once daily orally
  Arms: PAZOPANIB
Drug: Placebo — matching placebo 800 mg once daily orally
  Arms: PLACEBO

SUMMARY:
A randomized double blind phase III trial of Pazopanib versus placebo in patients with soft tissue sarcoma whose disease has progressed during or following prior therapy

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* High or intermediate grade of soft tissue sarcoma; Low grade tumours allowed provided there is disease progression.
* Metastatic and measurable disease (RECIST);
* Subjects can have received maximum of 4 prior lines of systemic therapies (including up to 2 combination regimens) for advanced disease. (Neo) adjuvant/maintenance treatments are not counted for this criterion;
* Last dose of prior therapy can be given upto 14 days prior to start of study if all ongoing toxicity from prior anticancer therapy are grade 1 or resolved (except alopecia).
* Must have failed anthracycline-based therapy and available standard chemotherapies at the treating institution except if medically contraindicated or refused by patient;
* No treatment with anti-angiogenesis inhibitors;
* Age > 18 years
* WHO PS 0-1;
* No leptomeningeal or brain metastases, normal bone marrow, liver, renal and cardiac functions;
* No prior history of malignancies other than sarcoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix or breast or the patient has been free of any other malignancies for > 3 years)
* Adequate bone marrow function; adequate blood clotting results; adequate hepatic and renal function;
* No poorly controlled hypertension;
* Clinically normal cardiac function;
* No clinically significant gastrointestinal abnormalities including malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* No cerebrovascular accidents 1
* No transient ischemic attack, deep vein thrombosis or pulmonary embolism within past six months;
* No active bleeding or bleeding diathesis;
* No hemoptysis within six weeks of study drug;
* No major surgery or trauma within 28 days of therapy treatment;
* Concomitant medication restriction;
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib
* Ability to swallow & retain oral medication
* Adequate contraception must be used;
* No Psychological familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before randomization in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (73):
- United States (9):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Clevand, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
- Australia (6):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Kurralta Park, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- GSK Investigational Site, Herlev, Denmark
- France (8):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Villejuif
- Germany (8):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Bad Saarow, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
- Italy (7):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Candiolo (TO), Piedmont
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Terni, Umbria
- Japan (8):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (5):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Valencia
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
- United Kingdom (6):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Background] van der Graaf WT, Blay JY, Chawla SP, Kim DW, Bui-Nguyen B, Casali PG, Schoffski P, Aglietta M, Staddon AP, Beppu Y, Le Cesne A, Gelderblom H, Judson IR, Araki N, Ouali M, Marreaud S, Hodge R, Dewji MR, Coens C, Demetri GD, Fletcher CD, Dei Tos AP, Hohenberger P; EORTC Soft Tissue and Bone Sarcoma Group; PALETTE study group. Pazopanib for metastatic soft-tissue sarcoma (PALETTE): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2012 May 19;379(9829):1879-86. doi: 10.1016/S0140-6736(12)60651-5. Epub 2012 May 16. PMID 22595799
- [Derived] Cesne AL, Bauer S, Demetri GD, Han G, Dezzani L, Ahmad Q, Blay JY, Judson I, Schoffski P, Aglietta M, Hohenberger P, Gelderblom H. Safety and efficacy of Pazopanib in advanced soft tissue sarcoma: PALETTE (EORTC 62072) subgroup analyses. BMC Cancer. 2019 Aug 13;19(1):794. doi: 10.1186/s12885-019-5988-3. PMID 31409302
- [Derived] Kawai A, Araki N, Hiraga H, Sugiura H, Matsumine A, Ozaki T, Ueda T, Ishii T, Esaki T, Machida M, Fukasawa N. A randomized, double-blind, placebo-controlled, Phase III study of pazopanib in patients with soft tissue sarcoma: results from the Japanese subgroup. Jpn J Clin Oncol. 2016 Mar;46(3):248-53. doi: 10.1093/jjco/hyv184. Epub 2016 Feb 10. PMID 26864131
- [Derived] Kasper B, Sleijfer S, Litiere S, Marreaud S, Verweij J, Hodge RA, Bauer S, Kerst JM, van der Graaf WTA. Long-term responders and survivors on pazopanib for advanced soft tissue sarcomas: subanalysis of two European Organisation for Research and Treatment of Cancer (EORTC) clinical trials 62043 and 62072. Ann Oncol. 2014 Mar;25(3):719-724. doi: 10.1093/annonc/mdt586. Epub 2014 Feb 6. PMID 24504442

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablets administered orally once daily for a duration until participants experienced disease progression, death, unacceptable toxicity, or participants withdrew consent
- Pazopanib: Pazopanib 200 milligrams (mg) and 400 mg film-coated tablets (containing pazopanib monohydrochloride) administered orally at a dose of 800 mg once daily for a duration until participants experienced disease progression, death, unacceptable toxicity, or participants withdrew consent
Period: Overall Study
Arm/Group | Placebo | Pazopanib
Started | 123 | 246
Ongoing - in Follow-up | 15 | 31
Completed | 0 | 0
Not Completed | 123 | 246
Not completed — Death | 102 | 203
Not completed — Missing | 4 | 9
Not completed — Participant Withdrew Consent | 2 | 2
Not completed — Ongoing - in Follow-up | 15 | 31
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pazopanib | Total
Number analyzed (Participants) | 123 | 246 | 369
Age Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (13.77) | 54.0 (14.92) | 53.2 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 147 | 216
  Male | 54 | 99 | 153
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 2 | 4 | 6
  American Indian or Alaska Native | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 2 | 0 | 2
  Asian - East Asian Heritage | 7 | 24 | 31
  Asian - Japanese Heritage | 16 | 31 | 47
  Asian - South East Asian Heritage | 2 | 2 | 4
  White - Arabic/North African Heritage | 2 | 1 | 3
  White - White/Caucasian/European Heritage | 89 | 174 | 263
  Mixed Race | 1 | 0 | 1
  Unknown | 2 | 9 | 11
Number of participants in the indicated soft tissue sarcoma (STS) subgroups at Baseline [Number; unit: participants] — Participants were categorized in the following histology subgroups of STS (as per the World Health Organization [WHO] classification, 2008): leiomyosarcoma, defined as malignant cancer of smooth muscle; synovial sarcoma, defined as cancer near the joints of the arm or leg; and other STS, defined as sarcoma without the tumor type of leiomyosarcoma or synovial sarcoma.
  participants
    Leiomyosarcoma | 49 | 109 | 158
    Synovial sarcoma | 13 | 25 | 38
    Other STS histologies | 61 | 112 | 173

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time interval between the date of randomization and the earliest date of either disease progression or death due to any cause. The diagnosis of progression was based on tumor measurements, according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 criteria, by independent radiologic assessment. The Kaplan-Meier method was used for PFS estimates.
Time Frame: From the date of randomization until the date of the first documented radiological progression or date of death from any cause, whichever came first (assessed for an average of 10 months)
Population: Intent-to-Treat (ITT) Population: all randomized participants analyzed in the treatment arm they were allocated by randomization.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 123 | 246
weeks | 7.0 [4.4 to 8.1] | 20.0 [17.9 to 21.3]
Statistical Analysis 1: Comparison: Placebo vs Pazopanib; Test type: Superiority or Other; p < 0.001, Log Rank — Stratified two-sided log rank p-value; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.26 to 0.48] — The HR was adjusted for World Health Organization (WHO) performance status scale (0 versus 1 at Baseline) and number of prior lines of systemic treatment for advanced disease (0/1 versus 2+)

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. The length of this interval was calculated as the date of death minus the date of randomization plus 1 day. Participants who were alive at the time of analysis were censored at the date of last follow-up. The interim OS analysis was conducted when 215 (77 percent [%]) of the 279 required death events had occurred in the study. The Kaplan-Meier method was used for OS estimates.
Time Frame: From the date of randomization until 215 deaths (assessed for an average of 12 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 123 | 246
months | 10.7 [9.0 to 13.1] | 12.6 [10.9 to 14.9]
Statistical Analysis 1: Comparison: Placebo vs Pazopanib; Test type: Superiority or Other; p = 0.256, Log Rank — Stratified two-sided log rank p-value; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.67 to 1.12] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants in the Indicated Categories for Overall Response Assessed by an Independent Radiologist and the Investigator
Description: Overall response is defined as the number of participants who had a complete response (CR) or a partial response (PR). According to RECIST, Version 1.0: CR, disappearance of all lesions; PR, a >=30% decrease in the sum of the longest dimensions (LD) of the target lesions (TLs) taking as a reference the baseline sum LD; Progressive disease (PD), a >=20% increase in the sum of the LD of TLs, or the appearance of >=1 new lesion; Stable Disease (SD), neither PR nor PD, persistence of >=1 non-TL. Participants with no follow-up radiological disease assessment were categorized as not evaluable (NE).
Time Frame: From the start of treatment until disease progression (assessed for an average of 10 months)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 123 | 246
participants
  CR, Independent radiologist assessed | 0 | 0
  PR, Independent radiologist assessed | 0 | 11
  SD, Independent radiologist assessed | 33 | 134
  PD, Independent radiologist assessed | 76 | 66
  NE, Independent radiologist assessed | 14 | 35
  CR, Investigator assessed | 0 | 0
  PR, Investigator assessed | 0 | 23
  SD, Investigator assessed | 36 | 138
  PD, Investigator assessed | 83 | 70
  NE, Investigator assessed | 4 | 15

4. Secondary Outcome: Time to Response Assessed by an Independent Radiologist and the Investigator
Description: Time to response was defined as the time from the date of randomization until the date of first documented evidence of CR or PR (whichever status was recorded first). The Kaplan-Meier method was used for time to response estimates.
Time Frame: From the date of randomization until the date of the first documented evidence of CR or PR (assessed for an average of 10 months)
Population: ITT Population. Only participants who achieved a confirmed CR or PR, as determined independently by the Independent Radiologist and the Investigator, were analyzed. Only results for the pazopanib arm are given because there was no response in the placebo arm.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 0 | 23
weeks
  Independent radiologist assessed, n=0, 11 |  | 8.4 [4.7 to 19.1]
  Investigator assessed, n=0, 23 |  | 8.1 [4.6 to 11.7]

5. Secondary Outcome: Duration of Response Assessed by the Independent Radiologist and the Investigator
Description: Duration of response was defined as the time from the date of the first documented evidence of CR or PR until the date of either the first documented sign of PD or death due to any cause. Participants who neither died nor progressed were censored at the date of the last adequate radiologic assessment. The Kaplan-Meier method was used for duration of response estimates.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 0 | 23
weeks
  Independent radiologist assessed, n=0, 11 |  | 38.9 [16.7 to 40.0]
  Investigator assessed, n=0, 23 |  | 32.1 [22.6 to 44.0]

6. Secondary Outcome: PFS in the Indicated Histology Subgroups of Soft Tissue Sarcoma (STS)
Description: PFS was defined as the time interval between the date of randomization and the earliest date of either disease progression or death due to any cause. Participants were analyzed for PFS in histology subgroups of STS (as per the World Health Organization [WHO] classification, 2008): leiomyosarcoma (malignant cancer of smooth muscle), synovial sarcoma (cancer near the joints of the arm or leg), and other STS (without the tumor type of leiomyosarcoma or synovial sarcoma), based on independent review.The Kaplan-Meier method was used for PFS estimates.
Time Frame: From the date of randomization until the date of the first documented progression or the date of death from any cause, whichever came first (assessed for an average of 10 months)
Population: ITT Population. The "n"s in the category titles represent the number of participants in each treatment arm with the indicated STS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 123 | 246
weeks
  Leiomyosarcoma, n=49, 109 | 8.1 [7.6 to 9.3] | 20.1 [13.3 to 23.1]
  Synovial sarcoma, n=13, 25 | 4.1 [3.7 to 8.9] | 17.9 [8.9 to 27.1]
  Other STS, n=61, 112 | 4.3 [4.0 to 7.9] | 20.1 [13.0 to 27.1]
Statistical Analysis 1: Comparison: Placebo vs Pazopanib; Test type: Superiority or Other; p < 0.001, Log Rank — Stratified two-sided log rank p-value for leiomyosarcoma; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.23 to 0.60] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Pazopanib; Test type: Superiority or Other; p = 0.005, Log Rank — Stratified two-sided log rank p-value for synovial sarcoma; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.19 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Pazopanib; Test type: Superiority or Other; p < 0.001, Log Rank — Stratified two-sided log rank p-value for other STS histologies; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.25 to 0.60] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from baseline in on-therapy SBP and DBP was calculated as the values at the indicated time points (Day 8 and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 88, 96, and 104) minus the value at baseline.
Time Frame: Baseline, Day 8, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 88, 96, and 104
Population: Safety Population: all participants who had started their allocated treatment (at least one dose of the study drug). Data were analyzed for participants who were on-therapy and provided data at the indicated time point.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 120 | 235
Millimeters of mercury
  SBP, Day 8, n=120, 235 | -0.6 (13.37) | 10.3 (15.96)
  SBP, Week 4, n=106, 224 | -0.2 (12.83) | 10.9 (19.47)
  SBP, Week 8, n=71, 180 | 0.0 (13.60) | 7.2 (17.46)
  SBP, Week 12, n=31, 115 | -3.1 (15.82) | 4.9 (18.21)
  SBP, Week 16, n=35, 136 | -0.6 (15.91) | 4.9 (18.49)
  SBP, Week 20, n=14, 66 | -2.6 (14.89) | 3.9 (19.84)
  SBP, Week 24, n=22, 107 | -3.8 (16.71) | 2.7 (20.24)
  SBP, Week 28, n=9, 41 | 0.2 (22.82) | 0.9 (15.70)
  SBP, Week 32, n=12, 76 | 2.8 (12.50) | 3.2 (18.89)
  SBP, Week 36, n=5, 24 | 3.6 (10.71) | 1.9 (17.71)
  SBP, Week 40, n=5, 62 | 6.8 (15.47) | 3.2 (19.75)
  SBP, Week 44, n=3, 16 | 6.0 (19.31) | 1.2 (19.45)
  SBP, Week 48, n=3, 37 | -1.7 (14.05) | -1.7 (16.90)
  SBP, Week 52, n=1, 6 | -4.0 (0) | 9.8 (18.28)
  SBP, Week 56, n=1, 27 | 16.0 (0) | 1.4 (20.86)
  SBP, Week 60, n=0, 6 | 0 (0) | 7.0 (18.60)
  SBP, Week 64, n=1, 15 | 20.0 (0) | -3.0 (19.26)
  SBP, Week 68, n=0, 2 | 0 (0) | 14.5 (3.54)
  SBP, Week 72, n=1, 9 | 8.0 (0) | -1.1 (15.83)
  SBP, Week 76, n=0, 1 | 0 (0) | 16.0 (0)
  SBP, Week 80, n=1, 5 | 19.0 (0) | -0.9 (22.66)
  SBP, Week 88, n=1, 3 | 3.0 (0) | 3.9 (22.90)
  SBP, Week 96, n=1, 2 | 13.0 (0) | -3.0 (14.14)
  SBP, Week 104, n=1, 1 | 18.0 (0) | 6.0 (0)
  DBP, Day 8, n=120, 235 | -0.2 (9.53) | 7.2 (10.68)
  DBP, Week 4, n=106, 224 | -0.2 (9.51) | 8.2 (11.37)
  DBP, Week 8, n=71, 180 | -0.3 (9.24) | 6.6 (12.18)
  DBP, Week 12, n=31, 115 | -0.1 (10.81) | 3.9 (11.31)
  DBP, Week 16, n=35, 136 | 0.8 (10.46) | 5.3 (12.12)
  DBP, Week 20, n=14, 66 | -0.3 (8.61) | 4.5 (12.22)
  DBP, Week 24, n=22, 107 | -1.6 (11.78) | 3.7 (14.44)
  DBP, Week 28, n=9, 41 | -1.9 (12.33) | 3.7 (11.28)
  DBP, Week 32, n=12, 76 | -2.0 (7.30) | 3.9 (11.59)
  DBP, Week 36, n=5, 24 | -6.6 (9.63) | 4.1 (13.28)
  DBP, Week 40, n=5, 62 | 3.4 (9.24) | 2.9 (13.34)
  DBP, Week 44, n=3, 16 | 4.7 (5.03) | 1.7 (12.48)
  DBP, Week 48, n=3, 37 | 2.0 (4.36) | 3.7 (12.01)
  DBP, Week 52, n=1, 6 | 1.0 (0) | 12.0 (15.06)
  DBP, Week 56, n=1, 27 | 12.0 (0) | 4.4 (12.28)
  DBP, Week 60, n=0, 6 | 0 (0) | 12.7 (14.39)
  DBP, Week 64, n=1, 15 | 10.0 (0) | -2.2 (14.21)
  DBP, Week 68, n=0, 2 | 0 (0) | 17.0 (25.46)
  DBP, Week 72, n=1, 9 | 13.0 (0) | 0.8 (12.88)
  DBP, Week 76, n=0, 1 | 0 (0) | 4.0 (0)
  DBP, Week 80, n=1, 5 | 14.0 (0) | -3.3 (15.15)
  DBP, Week 88, n=1, 3 | 9.0 (0) | 5.2 (3.87)
  DBP, Week 96, n=1, 2 | 6.0 (0) | 7.0 (5.66)
  DBP, Week 104, n=1, 1 | 12.0 (0) | 12.0 (0)

8. Secondary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline in on-therapy heart rate was calculated as the value at the indicated time points (Day 8 and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 88, 96, and 104) minus the value at baseline.
Time Frame: Baseline, Day 8, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 88, 96, and 104
Population: Safety Population. Data were analyzed for participants who were on-therapy and provided data at the indicated time point.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 113 | 225
beats per minute
  Day 8, n=113, 225 | 1.6 (12.61) | -4.4 (11.24)
  Week 4, n=98, 208 | 3.1 (13.06) | -2.7 (13.51)
  Week 8, n=66, 171 | 2.1 (15.03) | -1.6 (14.31)
  Week 12, n=29, 103 | 1.1 (17.32) | -2.4 (11.67)
  Week 16, n=31, 127 | 6.0 (16.78) | -3.7 (12.76)
  Week 20, n=12, 57 | 0.6 (22.95) | -3.4 (11.71)
  Week 24, n=21, 94 | 4.5 (18.14) | -5.0 (12.83)
  Week 28, n=7, 37 | -1.1 (27.99) | -3.8 (13.68)
  Week 32, n=12, 72 | -1.7 (18.38) | -2.7 (12.63)
  Week 36, n=5, 24 | -11.8 (32.57) | 0.9 (13.37)
  Week 40, n=5, 58 | -8.2 (30.19) | -2.4 (12.84)
  Week 44, n=3, 15 | 7.0 (16.09) | -0.9 (14.02)
  Week 48, n=3, 33 | 9.0 (18.00) | 1.9 (14.38)
  Week 52, n=1, 5 | -8.0 (0) | -3.4 (16.96)
  Week 56, n=1, 24 | 31.0 (0) | -0.4 (15.14)
  Week 60, n=0, 6 | 0 (0) | 4.3 (15.13)
  Week 64, n=1, 13 | 36.0 (0) | -1.5 (13.56)
  Week 68, n=0, 2 | 0 (0) | 9.5 (0.71)
  Week 72, n=1, 8 | 14.0 (0) | 2.6 (12.60)
  Week 76, n=0, 1 | 0 (0) | 5.0 (0)
  Week 80, n=1, 5 | 24.0 (0) | 2.8 (16.08)
  Week 88, n=1, 3 | 9.0 (0) | -3.0 (10.58)
  Week 96, n=1, 2 | 17.0 (0) | -5.0 (4.24)
  Week 104, n=1, 1 | 30.0 (0) | 1.0 (0)

9. Secondary Outcome: Number of Participants With the Indicated Grade Shifts From Baseline Grade for Hemoglobin Level, Lymphocyte Count, White Blood Cell Count, Neutrophil Count, and Platelet Count
Description: Shifts in hematology values by grade were summarized based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE Version 3.0). Grade refers to the severity of the AE. The CTCAE Version 3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline. Participants with a missing baseline grade were assumed to have a baseline Grade of 0. Any increase in grade from baseline and shifts to Grade 3 (severe AE) and 4 (life-threatening or disabling AE) at any point in the study after baseline are reported.
Time Frame: From baseline (Day 1) until study drug discontinuation or end of treatment (assessed for an average of 20 weeks)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 123 | 239
participants
  Hemoglobin, Any Increase, n=123, 239 | 28 | 65
  Hemoglobin, Increase to Grade 3, n=123, 239 | 1 | 11
  Hemoglobin, Increase to Grade 4, n=123, 239 | 1 | 4
  Lymphocytes, Any Increase, n=123, 238 | 44 | 102
  Lymphocytes, Increase to Grade 3, n=123, 238 | 11 | 23
  Lymphocytes, Increase to Grade 4, n=123, 238 | 2 | 0
  Neutrophils, Any Increase, n=123, 239 | 8 | 79
  Neutrophils, Increase to Grade 3, n=123, 239 | 0 | 10
  Neutrophils, Increase to Grade 4, n=123, 239 | 0 | 0
  Platelets, Any Increase, n=123, 239 | 7 | 86
  Platelets, Increase to Grade 3, n=123, 239 | 0 | 7
  Platelets, Increase to Grade 4, n=123, 239 | 0 | 2
  White Blood Cells, Any Increase, n=123, 239 | 18 | 106
  White Blood Cells, Increase to Grade 3, n=123, 239 | 0 | 3
  White Blood Cells, Increase to Grade , n=123, 239 | 0 | 0

10. Secondary Outcome: Number of Participants With the Indicated Grade Shifts From Baseline Grade for Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Albumin, Creatinine, Hyper/Hypoglycemia, Hyper/Hypokalemia, Hyper/Hyponatremia, and Total Bilirubin
Description: Shifts in clinical chemistry values by grade were summarized based on the NCI CTCAE Version 3.0. Participants with a missing baseline grade were assumed to have a baseline Grade of 0. Any increase in grade from baseline and shifts to Grade 3 and 4 at any point in the study after baseline are reported. alkaline phosphatase, ALKP; alanine aminotransferase, ALT; aspartate aminotransferase, AST. Hyper/hypoglycemia refers to high/low glucose; hyper/hypokalemia refers to high/low potassium; hyper/hyponatremia refers to high/low sodium.
Time Frame: From baseline (Day 1) until study drug discontinuation or end of treatment (assessed for an average of 20 weeks)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 123 | 239
participants
  ALKP, Any Increase, n=123, 237 | 28 | 77
  ALKP, Increase to Grade 3, n=123, 237 | 1 | 7
  ALKP, Increase to Grade 4, n=123, 237 | 0 | 0
  ALT, Any Increase, n=123, 237 | 22 | 110
  ALT, Increase to Grade 3, n=123, 237 | 3 | 18
  ALT, Increase to Grade 4, n=123, 237 | 1 | 5
  AST, Any Increase, n=123, 239 | 27 | 122
  AST, Increase to Grade 3, n=123, 239 | 2 | 13
  AST, Increase to Grade 4, n=123, 239 | 0 | 6
  Albumin, Any Increase, n=123, 239 | 26 | 81
  Albumin, Increase to Grade 3, n=123, 239 | 0 | 2
  Albumin, Increase to Grade 4, n=123, 239 | 0 | 0
  Creatinine, Any Increase, n=123, 239 | 9 | 28
  Creatinine, Increase to Grade 3, n=123, 239 | 0 | 1
  Creatinine, Increase to Grade 4, n=123, 239 | 0 | 0
  Hyperglycemia, Any Increase, n=122, 238 | 43 | 106
  Hyperglycemia, Increase to Grade 3, n=122, 238 | 2 | 1
  Hyperglycemia, Increase to Grade 4, n=122, 238 | 0 | 0
  Hyperkalemia, Any Increase, n=123, 238 | 13 | 37
  Hyperkalemia, Increase to Grade 3, n=123, 238 | 0 | 3
  Hyperkalemia, Increase to Grade 4, n=123, 238 | 0 | 0
  Hypernatremia, Any Increase, n=123, 238 | 3 | 10
  Hypernatremia, Increase to Grade 3, n=123, 238 | 0 | 0
  Hypernatremia, Increase to Grade 4, n=123, 238 | 0 | 0
  Hypoglycemia, Any Increase, n=122, 238 | 4 | 21
  Hypoglycemia, Increase to Grade 3, n=122, 238 | 0 | 1
  Hypoglycemia, Increase to Grade 4, n=122, 238 | 0 | 0
  Hypokalemia, Any Increase, n=123, 238 | 11 | 32
  Hypokalemia, Increase to Grade 3, n=123, 238 | 1 | 6
  Hypokalemia, Increase to Grade 4, n=123, 238 | 0 | 1
  Hyponatremia, Any Increase, n=123, 238 | 25 | 74
  Hyponatremia, Increase to Grade 3, n=123, 238 | 4 | 9
  Hyponatremia, Increase to Grade 4, n=123, 238 | 0 | 0
  Total Bilirubin, Any Increase, n=122, 237 | 9 | 68
  Total Bilirubin, Increase to Grade 3, n=122, 237 | 2 | 3
  Total Bilirubin, Increase to Grade 4, n=122, 237 | 0 | 0

11. Secondary Outcome: Number of Participants With the Indicated Absolute Percent Change From Baseline (BL) in Left Ventricular Ejection Fraction (LVEF) at Any Time Post-BL (Worst Case On-therapy)
Description: LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction and is used to determine cardiac function (based on the institutional lower limit of normal [LLN]). LVEF was assessed at BL, Week 12, and every second scheduled visit thereafter until study drug discontinuation and end of treatment or as clinically indicated by using multi-gated acquisition scan (MUGA) or echocardiogram (ECHO). Absolute change from BL was calculated as the on-study value minus the baseline value (LVEF is calculated as a percentage).
Time Frame: Baseline (within 14 days of the first dose of study drug) and any time post-baseline until study drug discontinuation or end of treatment (assessed for an average of 20 weeks)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib
Number analyzed (Participants) | 39 | 140
participants
  Any Increase | 15 | 39
  No Change | 6 | 14
  0 to <10% Decrease | 15 | 66
  10 to 19% Decrease | 3 | 15
  >=20% Decrease | 0 | 6
  >=10% Decrease and >= LLN | 3 | 8
  >=10% Decrease and below LLN | 0 | 13
  >=20% Decrease and >= LLN | 0 | 1
  >=20% Decrease and below LLN | 0 | 5

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Baseline through End of Study (average of 20 study weeks).
Description: The Safety Population, comprised of all participants who had started their allocated treatment (at least one dose of the study drug), was used for all safety analyses.
Arm/Group | Placebo | Pazopanib
Serious Adverse Events (participants affected / at risk) | 29/123 | 99/240
Other Adverse Events (participants affected / at risk) | 108/123 | 232/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=123) | Pazopanib (N=240)
Alanine aminotransferase increased (Investigations) | 1 | 9
Hemoglobin decreased (Investigations) | 2 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 6
Gamma-glutamyltransferase increased (Investigations) | 0 | 6
Platelet count decreased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 2
Neutrophil percentage (Investigations) | 1 | 2
Alanine aminotransferase (Investigations) | 1 | 1
Aspartate aminotransferase (Investigations) | 0 | 2
Blood potassium decreased (Investigations) | 1 | 1
Lymphocyte percentage (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 2
Bilirubin conjugated (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood cholesterol abnormal (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Hemoglobin (Investigations) | 0 | 1
Neutrophil percentage decreased (Investigations) | 0 | 1
Urine protein/creatinine ratio (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 1 | 2
Abscess (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 1
Lactobacillus infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 4
Colonic obstruction (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Hematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Peritoneal hemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 5
Chest pain (General disorders) | 0 | 4
Pyrexia (General disorders) | 3 | 1
Performance status decreased (General disorders) | 0 | 3
Disease progression (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Localized edema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 2 | 6
Hemorrhage (Vascular disorders) | 0 | 1
Ischemia (Vascular disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Hemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Mass (General disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=123) | Pazopanib (N=240)
Nausea (Gastrointestinal disorders) | 27 | 135
Diarrhea (Gastrointestinal disorders) | 19 | 141
Vomiting (Gastrointestinal disorders) | 14 | 81
Gastrointestinal pain (Gastrointestinal disorders) | 11 | 57
Constipation (Gastrointestinal disorders) | 21 | 39
Stomatitis (Gastrointestinal disorders) | 4 | 27
Abdominal pain upper (Gastrointestinal disorders) | 7 | 19
Dry mouth (Gastrointestinal disorders) | 6 | 16
Dyspepsia (Gastrointestinal disorders) | 2 | 18
Fatigue (General disorders) | 59 | 157
Edema peripheral (General disorders) | 11 | 33
Pyrexia (General disorders) | 12 | 25
Chest pain (General disorders) | 7 | 26
Chills (General disorders) | 1 | 14
Weight decreased (Investigations) | 9 | 122
Ear, nose and throat examination abnormal (Investigations) | 3 | 29
Weight increased (Investigations) | 9 | 12
Hair color changes (Skin and subcutaneous tissue disorders) | 3 | 93
Exfoliative rash (Skin and subcutaneous tissue disorders) | 11 | 46
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 29
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 28
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 16
Dysgeusia (Nervous system disorders) | 4 | 66
Headache (Nervous system disorders) | 10 | 57
Dizziness (Nervous system disorders) | 5 | 26
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 56
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 56
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 43
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 19
Decreased appetite (Metabolism and nutrition disorders) | 23 | 97
Hypertension (Vascular disorders) | 7 | 101
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 71
Insomnia (Psychiatric disorders) | 7 | 24
Anxiety (Psychiatric disorders) | 8 | 20
Left ventricular dysfunction (Cardiac disorders) | 5 | 19
Hypothyroidism (Endocrine disorders) | 0 | 20
Nasopharyngitis (Infections and infestations) | 7 | 13
Vision blurred (Eye disorders) | 2 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.